CLINICAL TRIAL: NCT02093429
Title: A Randomized, Open-Label, 2-Stage Study of INCB047986 Administered Orally to Subjects With Primary Myelodysplastic Syndrome (MDS) Refractory to or Unlikely to Respond to Erythropoiesis-Stimulating Agents (ESAs)
Brief Title: Randomized Open-Label Study of INCB047986 in Subjects With Primary Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 47986-201
Record Dates: First submitted 2014-01-03; First posted 2014-03-21 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: MDS (Myelodysplastic Syndrome)
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- INCB047986 4 mg (Experimental): Participants will receive INCB047986 4 mg once daily for at least 16 weeks.
  Interventions: Drug: INCB047986
- INCB047986 6 mg (Experimental): Participants will receive INCB047986 6 mg once daily for at least 16 weeks.
  Interventions: Drug: INCB047986
- INCB047986 10 mg (Experimental): Participants will receive INCB047986 10 mg once daily for at least 16 weeks.
  Interventions: Drug: INCB047986

INTERVENTIONS:
Drug: INCB047986 — INCB047986 will be supplied as tablets.

SUMMARY:
The study design includes a 3-dose randomization phase to determine effective doses of INCB047986 in patients with myelodysplastic syndrome (MDS) who are refractory or unlikely to respond to erythropoiesis-stimulating agents (ESAs) followed by an extension phase.

DETAILED DESCRIPTION:
After 50% of the subjects have completed 16 weeks of treatment (10 subjects in each dose group), a planned interim analysis will be conducted to determine which, if any, dose levels warrant further investigation based on observing at least 3 responses for hematologic improvement in erythrocytes (HI-E) and adequate safety and tolerability.

Subjects who do not meet the response criteria for erythroid improvement may be treated with ESA in combination with INCB047986 for an additional 16 weeks.

The study comprises:

Screening: up to 4 weeks. Treatment Phase 1: at least 16 weeks of INCB047986. Treatment Phase 2: at least 8 and up to 16 weeks of INCB047986 in combination with ESA if failed treatment in Phase 1.

Extension Phase: Subjects receiving benefit from either therapy may continue indefinitely or until the study is terminated.

Follow-Up: 30 (± 7) days after the last dose of INCB047986 is taken.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older.
* Subjects must be diagnosed with MDS according to the World Health Organization (WHO) classification for de novo or primary MDS (Vardiman et al 2009).
* Subjects who require RBC transfusions or are either refractory to or unlikely to respond to ESA therapy should meet one of the following criteria:

  * ESA failure as defined by no improvement in Hgb of at least 1.5 g/dL after 8 weeks of at least 40,000 IU per week of EPO (or equivalent).
  * Have a serum erythropoietin (EPO) of ≥ 500 IU and Hgb level < 10.0 g/dL.
  * Transfusion dependence defined as requiring at least 4 units of packed red blood cells (RBCs) for a Hgb of < 9 g/dL over the 8 weeks prior to screening.
* Subjects may not have received hypomethylating agents or immunosuppressive therapy for their MDS prior to this study.

Exclusion Criteria:

* Subjects at high risk for transformation to acute leukemia as evidenced by poor karyotype or peripheral blood blasts > 10%.
* Subjects with severely compromised bone marrow function as evidenced by trilineage cytopenias with anemia (Hgb < 10 g/L, platelets < 100 × 109/L, and absolute neutrophil count (ANC) < 1.8 × 109/L).
* Subjects who harbor the 5q deletion chromosomal aberration.
* Subjects with chronic myelomonocytic leukemia (CMML).
* Women who are pregnant or breastfeeding, and men and women who cannot comply with requirements to avoid fathering a child or becoming pregnant, respectively.
* Subjects with impaired liver function, end stage renal disease on dialysis, or clinically significant concurrent infections requiring therapy.
* Subjects with unstable cardiac function.
* Invasive malignancies over the previous 2 years except treated basal or squamous carcinomas of the skin, completely resected intraepithelial carcinoma of the cervix, Stage 1 or 2 treated prostate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a response for Hematologic Improvement in Erythrocytes (HI-E) during any 8-week period within the first 16-week treatment period with INCB047986 Monotherapy. | Baseline to Week 16
Safety and tolerability of INCB047986 as assessed by summary of clinical laboratory assessments and summary of Adverse Events (AEs). | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William V. Williams, M.D., Study Director — Incyte Corporation
Locations (7):
- United States (7):
  - Highland, California
  - Indianapolis, Indiana
  - Morristown, New Jersey
  - Somerville, New Jersey
  - Germantown, Tennessee
  - Houston, Texas
  - Burlington, Vermont